CLINICAL TRIAL: NCT07319611
Title: Investigation of the Effects of High-Intensity Interval Exercise and Moderate-Intensity Continuous Exercise on Limb Volume, Functional Capacity, and Quality of Life in Patients With Lipedema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MarmaraU-FTR-GNY-01
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Lipedema; Exercise Therapy; High Intensity Interval Training
Keywords: lipedema; high intensity interval training; moderate intensity continuous training
MeSH Terms: conditions — Lipedema | interventions — Intermittent Pneumatic Compression Devices; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Pneumatic Compression + Home-Based Walking Program (Experimental): Participants in this group will receive 15 sessions of intermittent pneumatic compression (IPC) therapy combined with a home-based walking program for 10 weeks. IPC will be applied 3 times per week at 50 mmHg pressure for 30 minutes using the DoctorLife LX7 Max device. Participants will also be instructed to walk at least 10,000 steps daily, monitored via a validated pedometer mobile application (PACER). Exercise adherence will be supported through follow-up and exercise diaries.
  Interventions: Device: Intermittent Pneumatic Compression (IPC); Behavioral: Home-Based Walking Program
- Intermittent Pneumatic Compression + High-Intensity Interval Training (HIIT) (Experimental): This group will receive 15 sessions of IPC therapy and 30 sessions of supervised high-intensity interval training (HIIT) performed on a stationary cycle ergometer. The program will last 10 weeks (3 sessions per week). Each session will include a 5-minute warm-up, seven 1-minute high-intensity intervals (with 1-minute active recovery periods), and a 5-minute cool-down, for a total of 23 minutes. Exercise intensity will be individually determined using the Graded Cycling Test with Talk Test (GCT-TT), corresponding to Borg scale 14-16 for intervals. Participants will be continuously monitored for heart rate, rhythm, oxygen saturation, and blood pressure during exercise.
  Interventions: Device: Intermittent Pneumatic Compression (IPC); Behavioral: High-Intensity Interval Training (HIIT)
- Intermittent Pneumatic Compression + Moderate-Intensity Continuous Training (MICT) (Experimental): This group will receive 15 sessions of IPC therapy and 30 sessions of supervised moderate-intensity continuous training (MICT) over 10 weeks. Each session (55 minutes total) will consist of a 5-minute warm-up, 45 minutes of steady-state cycling at 50% of maximal power output (from the GCT-TT), and a 5-minute cool-down. The corresponding effort equates to Borg scale 12. Sessions will occur 3 times per week under physiotherapist supervision with continuous monitoring of vital signs.
  Interventions: Device: Intermittent Pneumatic Compression (IPC); Behavioral: Moderate-Intensity Continuous Training (MICT)

INTERVENTIONS:
Device: Intermittent Pneumatic Compression (IPC) — Applied to both lower limbs for 30 minutes at 50 mmHg, 3 times per week for 5 weeks using DoctorLife LX7 Max device. Used in all study arms.
Behavioral: Home-Based Walking Program — Participants perform ≥10,000 steps/day using PACER pedometer app; encouraged through exercise logs and follow-up.
  Arms: Intermittent Pneumatic Compression + Home-Based Walking Program
Behavioral: High-Intensity Interval Training (HIIT) — Supervised cycling-based interval exercise, 3×/week for 10 weeks, individualized by GCT-TT protocol.
  Arms: Intermittent Pneumatic Compression + High-Intensity Interval Training (HIIT)
Behavioral: Moderate-Intensity Continuous Training (MICT) — Supervised continuous cycling exercise, 3×/week for 10 weeks, at 50% GCT-TT power output.
  Arms: Intermittent Pneumatic Compression + Moderate-Intensity Continuous Training (MICT)

SUMMARY:
This randomized controlled clinical study aims to investigate and compare the effects of high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT), when combined with intermittent pneumatic compression (IPC) therapy, on limb volume, functional capacity, pain, fatigue, anxiety, depression, sleep quality, and quality of life in women with lipedema.

Lipedema is a chronic, progressive adipose tissue disorder primarily affecting women, characterized by abnormal and symmetrical fat accumulation in the lower extremities that does not improve with weight loss or limb elevation. It is often misdiagnosed as obesity or lymphedema, leading to delayed treatment. Lipedema causes pain, swelling, bruising, mobility limitation, and reduced quality of life.

Conservative treatment options include compression therapy, manual lymphatic drainage, and exercise. IPC is a non-invasive treatment used to reduce limb volume and pain while improving function and quality of life. Exercise is also a cornerstone of conservative management, but the optimal exercise intensity for lipedema remains unclear.

In this study, 69 female patients aged 18-65 years diagnosed with lipedema according to Halk and Damstra criteria will be randomly assigned into three groups:

IPC + Home-based walking program

IPC + High-Intensity Interval Training (HIIT)

IPC + Moderate-Intensity Continuous Training (MICT)

All participants will receive 15 IPC sessions (3 times per week for 5 weeks). The exercise programs (HIIT or MICT) will continue for 10 weeks, supervised by a physiotherapist. The home-based group will be encouraged to walk ≥10,000 steps daily using a pedometer application.

Primary outcome: Change in limb volume measured by circumferential measurements and the truncated cone formula.

Secondary outcomes: Pain (VAS), functional capacity (6-Minute Walk Test), muscle strength (dynamometry), pressure pain threshold (algometry), physical activity (IPAQ-SF), lower extremity function (LEFS), quality of life (SF-12), sleep quality (PSQI), fatigue (FSS), and anxiety/depression (HADS).

Measurements will be taken at baseline (T0), after 15 IPC sessions (T1), and after 30 total sessions or 10 weeks (T2).

The investigators hypothesize that both HIIT and MICT combined with IPC will provide superior improvements in physical and psychological outcomes compared to IPC with a home-based walking program alone.

DETAILED DESCRIPTION:
Detailed Description

This is a prospective, single-blind (assessor-blinded), randomized controlled trial conducted at Marmara University Pendik Training and Research Hospital, Department of Physical Medicine and Rehabilitation between November 2025 and November 2026.

The study will include 69 female participants diagnosed with lipedema according to clinical criteria. Participants will be randomly assigned (using www.randomizer.org) into three parallel groups (n=23 per group). Randomization and outcome assessment will be performed by independent evaluators blinded to group allocation.

Interventions

Intermittent Pneumatic Compression (IPC): 15 sessions, 3 times/week, using DoctorLife LX7 Max device at 50 mmHg for 30 minutes per session.

HIIT Group: 30 sessions, 3 times/week for 10 weeks, each lasting 23 minutes (5 min warm-up, 7 one-minute intervals with one-minute rests, and 5 min cool-down). Intensity determined by Graded Cycling Test with Talk Test (GCT-TT).

MICT Group: 30 sessions, 3 times/week for 10 weeks, each lasting 55 minutes (5 min warm-up, 45 min at 50% GCT-TT power, 5 min cool-down).

Home-based Walking Group: Encouraged to walk ≥10,000 steps daily using a validated pedometer app (PACER), supported by motivational follow-up and exercise diaries.

All exercise sessions will be supervised by a physiotherapist, and participants will be continuously monitored for heart rate, rhythm, oxygen saturation, and blood pressure.

Assessments

Measurements will include:

Limb volume (circumferential measurements every 8 cm, truncated cone formula)

6-Minute Walk Test (6MWT) for functional capacity

Isometric quadriceps strength using a hand-held dynamometer

Pressure pain threshold via algometer

VAS, LEFS, SF-12, PSQI, FSS, HADS, and IPAQ-SF questionnaires

Data collection will occur at three time points: baseline (T0), after 15 IPC sessions (T1), and at the end of 10 weeks (T2).

Statistical Plan

Power analysis (f=0.25, α=0.05, power=0.80) determined a total sample size of 57, increased to 69 to account for 20% dropout. Data will be analyzed using repeated measures ANOVA to compare time × group interactions.

Expected Outcomes

The study expects that both HIIT and MICT combined with IPC will significantly reduce limb volume and pain, and improve functional capacity, sleep, fatigue, and quality of life compared to home-based walking with IPC alone.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-65 years
* Able to read and write (literate)
* Clinically diagnosed with lipedema according to Halk and Damstra criteria

Exclusion Criteria:

* Pregnancy or breastfeeding
* Illiteracy
* Refusal or inability to provide written/signed consent
* Lower extremity fracture, trauma, or surgery within the past 12 months
* Cardiopulmonary diseases that contraindicate exercise participation
* Development of intolerance exercise sessions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Lower Extremity Volume (mL) | Baseline (Day 1), after 15 IPC sessions (Day 36), and post-intervention (Day 71)
  Lower limb volume will be calculated using circumferential measurements taken every 8 cm along both legs in the standing position. Volumetric values will be derived using the truncated cone formula. The primary endpoint is the change in total limb volume from baseline to week 10. Measurements will be conducted by a blinded assessor.

SECONDARY OUTCOMES:
Change in Functional Exercise Capacity (6-Minute Walk Test Distance, meters) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  The 6-Minute Walk Test measures the distance a participant can walk on a flat surface in six minutes. It reflects overall functional capacity and endurance. The change from baseline to week 10 will be compared between groups.
Change in Physical Activity Level (International Physical Activity Questionnaire-Short Form; MET-min/week) | Baseline (Day 0), and end of week 10 (Day 71)
  The IPAQ-SF assesses physical activity intensity and duration. Higher scores indicate greater activity level.
Change in Fatigue Severity (Fatigue Severity Scale, FSS; 9-63) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  The FSS measures the impact of fatigue on daily functioning. Scores ≥36 indicate severe fatigue. Lower post-treatment scores indicate improvement.
Change in Quality of Life (SF-12 Physical and Mental Composite Scores) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  The SF-12 questionnaire evaluates physical and mental components of quality of life. Higher scores represent better health-related quality of life.
Change in Lower Extremity Functional Scale (LEFS; 0-80) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  The LEFS assesses lower limb functional abilities. Each item is rated 0-4; total score ranges 0-80, with higher scores indicating better function.
Change in Pressure Pain Threshold (kg/cm²) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  Pressure pain threshold will be measured using a digital algometer on the lateral thigh and dorsum of the hand (reference point). Increased threshold values indicate improved pain tolerance.
Change in Isometric Quadriceps Strength (kgf) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  Maximal isometric knee extension strength will be measured bilaterally using an electronic hand-held dynamometer at 60° knee flexion. The average of two trials will be recorded. Higher values indicate greater strength.
Change in Pain Intensity (VAS; 0-100 mm) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  Pain intensity in both lower limbs will be assessed using a 100-mm Visual Analog Scale (VAS) under three conditions: movement, rest, and night pain. Higher scores indicate greater pain severity. The primary comparison is the change from baseline to week 10.
Change in Sleep Quality (Pittsburgh Sleep Quality Index, PSQI; 0-21) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  The PSQI assesses sleep quality; total score >5 indicates poor sleep. Lower scores represent better sleep quality.
Change in Anxiety and Depression (Hospital Anxiety and Depression Scale, HADS) | Baseline (Day 0), end of week 5 (Day 36), and end of week 10 (Day 71)
  HADS includes anxiety (HADS-A) and depression (HADS-D) subscales, each ranging from 0-21. Higher scores reflect more severe symptoms. Lower scores post-intervention indicate improvement.

OTHER OUTCOMES:
Adherence to Exercise and Treatment Program | Throughout the 10-week intervention period; summarized at post-intervention (Day 71)
  Measured as the percentage of attended exercise sessions (out of 30 planned) and mean daily step count from pedometer data in the home-based walking group. Used to assess adherence and compliance.
Adverse Events and Cardiovascular Safety | Throughout the 10-week intervention period; summarized at post-intervention (Day 71)
  Monitoring of adverse events during IPC or exercise sessions, including vital signs (heart rate, rhythm, oxygen saturation, and blood pressure) recorded each session.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz BAHAR ÖZDEMİR, Associate Professor, Study Director — Marmara University Pendik Training and Research Hospital
Locations (1):
- Marmara University Pendik Training and Research Hospital, Department of Physical Medicine and Rehabilitation, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this study, including demographic characteristics, outcome measures (e.g., limb volume, 6-minute walk distance, pain scores), and adverse event data, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available 6 months after publication of the main results and remain accessible for at least 5 years following publication.
Access Criteria: Qualified researchers may request access to the de-identified dataset and supporting documentation by submitting a brief research proposal and data access agreement to the corresponding investigator (Assoc. Prof. Dr. Yeliz Bahar Ozdemir, Marmara University, Istanbul, Turkey). Data will be shared via a secure institutional data repository upon approval by the principal investigator and the Marmara University Ethics Committee.
URL: https://www.marmara.edu.tr/